CLINICAL TRIAL: NCT00017355
Title: Mature Dendritic Cell Immunotherapy Of Metastatic Melanoma- A Phase I Trial
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor Health Care System (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068680; BAYUMC-000048; NCI-4170
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2003-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Filgrastim

INTERVENTIONS:
Biological: filgrastim
Biological: therapeutic autologous dendritic cells

SUMMARY:
RATIONALE: Vaccines made from a patient's white blood cells mixed with tumor antigens may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of antigen-pulsed dendritic cell vaccine in patients with metastatic melanoma.
* Determine the longevity of melanoma-specific immunity in patients treated with this regimen.
* Perform serial analysis of T-cell and B-cell function in patients treated with this regimen.

OUTLINE: Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily on days 1-6 or 1-7. Patients undergo apheresis on days 6 and 7 or 6-8 to obtain peripheral blood mononuclear cells (PBMC). PBMC are processed for CD34+ cell isolation. These autologous CD34+ hematopoietic progenitor cells are cultured to generate dendritic cells (DC). DC are then pulsed with endotoxin-free keyhole limpet hemocyanin and HLA-A2-01 restricted flu-matrix peptides derived from melanoma-associated tumor antigens (MART-1:27-35, gp100:209-217, and MAGE-3). Antigen-pulsed DC are incubated with interferon alfa to induce DC maturation.

Patients receive priming injections of antigen-pulsed DC vaccine SC once every 2 weeks for 8 weeks. Treatment repeats at 2, 3, 4, and 5 months after the last priming injection in the absence of unacceptable toxicity or disease progression.

Patients are followed at 2 and 4 weeks and then every 3 months for 1.5 years.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma
* HLA-A2-01 phenotype
* Measurable disease
* No active CNS or hepatic metastases

PATIENT CHARACTERISTICS:

Age:

* 21 and over

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* See Disease Characteristics
* No viral hepatitis

Renal:

* Not specified

Cardiovascular:

* No prior venous thrombosis, angina pectoris, or congestive heart failure
* Lactate dehydrogenase less than 2 times normal

Pulmonary:

* No prior asthma

Immunologic:

* Intradermal skin test positivity to mumps, Candida, or streptokinase antigen
* No known sensitivity to E. coli drug preparations
* No prior allergy to influenza vaccine
* No active infection
* No prior autoimmune disease (e.g., lupus erythematosus, rheumatoid arthritis, or thyroiditis)

Other:

* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 8 weeks since prior interleukin-2
* At least 4 weeks since prior interferon alfa

Chemotherapy:

* At least 8 weeks since prior chemotherapy

Endocrine therapy:

* At least 2 weeks since prior corticosteroids
* No concurrent corticosteroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent immunosuppressive agents
* At least 2 weeks since prior immunosuppressive agents

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W. Fay, MD, Study Chair — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States